CLINICAL TRIAL: NCT02596776
Title: Cold Induced Changes in Human Subcutaneous White Adipose
Brief Title: Cold Induced Changes in White Adipose
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Philip Kern (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Philip Kern, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15-0663; R01DK107646 (NIH)
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Obese; Normal Body Weight; Prediabetes; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Prediabetic State; Metabolic Syndrome | interventions — Propranolol; Deuterium Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fat biopsy (Active Comparator): From each abdominal and thigh biopsy, between 0.5 - 3 g of tissue is obtained (often less from the thigh), which is used for immunohistochemistry and frozen for subsequent RNA or protein isolation.
  Interventions: Procedure: Fat biopsy
- Propranolol and Fat Biopsy (Experimental): From each abdominal and thigh biopsy, tissue will be examined for gene expression, with a focus on genes believed to be involved in adipose beiging (PGC1α, UCP1, TMEM26, IL4, Metrnl, CPA3, Siglec 8, tyrosine hydroxylase, others), and with immunohistochemistry, with a focus on beige adipocytes, macrophages, eosinophils and mast cells.
  Interventions: Procedure: Fat biopsy; Drug: Propranolol and fat biopsy
- Heavy Water and Fat Biopsy (Active Comparator): The investigator will measure in vivo adipose lipolysis and triglyceride (TG) turnover in response to cold to physiologically demonstrate the impact of cold exposure on tissue function. The subjects will then be given 50 mL sterile containers of 70% 2H2O and consume two 50 mL vials per day during the remainder of the 5-week labeling period. Plasma and urine will be collected weekly so that body 2H2O can be measured.
  Interventions: Procedure: Fat biopsy; Other: heavy water and fat biopsy

INTERVENTIONS:
Procedure: Fat biopsy — up to 16 biopsy samples will be taken from each subject
Drug: Propranolol and fat biopsy — subset of subjects will receive propranolol and have fat biopsy performed
  Arms: Propranolol and Fat Biopsy
Other: heavy water and fat biopsy — subset of subjects will be given heavy water and have fat biopsy performed
  Arms: Heavy Water and Fat Biopsy

SUMMARY:
An adaptation to a cold environment is a tendency to generate heat within our body. Some of this heat comes from our fat tissue. Although most fat tissue is "white fat", there are pockets deep within the body that are called "brown fat", which are specially adapted to burning fat and making heat. The investigator believes that our white fat, just underneath the surface of our skin, also has this property to burn fat and make heat, although not at the high level of brown fat. This study is to examine this fat-burning property of the white fat under the skin in response to seasons and to cold. Many such studies have been done in mice, but little has been done in humans.

There are a number of factors, including age, weight, and medical history, that may make a person eligible or ineligible to participate in this study. Certain medications could make a person ineligible, but if these medications can be safely altered, the individual may become eligible.

DETAILED DESCRIPTION:
Metabolic syndrome is a condition involving elevated levels of fat in the blood, a tendency towards diabetes, hypertension, and too much fat around the abdomen (an increased waistline). Individuals with metabolic syndrome often have impaired glucose tolerance, which is a condition where blood sugar is normal before a person eats, but is too high after drinking a sugary drink. This is due to an abnormality in the body's sensitivity to insulin (insulin resistance), which is due in part to an inability of muscle to take up glucose. People with metabolic syndrome have inflammation in their fat tissue and this inflammation in the fat tissue may impair the ability of the white fat to burn fat and continue to promote obesity.

This study involves three arms. A propranolol with biopsy arm, a heavy water with biopsy arm, and a biopsy only arm. The goal is to understand the response of fat to cold, either acutely, or after repeated cold exposure, or in response to a change in seasons.

Individuals (subjects) accepted into the study will report to the UK Center for Clinical and Translational Science (CCTS) research unit for baseline testing and repeated procedures. Participants will then be asked to have the same procedures done approximately 6 months later.

Subjects enrolled into the study will need to come to the CCTS Unit for multiple visits. Most of these visits will be less than 1 hour, but 6 visits will involve procedures and will vary in time ranging from 4 hour to 6 hours. If a subject participates in all aspects of the study (fat biopsy from multiple depots, short term, long term, and seasons, then their total participation will be approximately 28 visits over 6-7 months. However, for most subjects, their participation will involve fewer visits, at the discretion of the principal investigator.

The first visit will involve the consent process, followed by baseline fasting blood samples and the oral glucose tolerance test. If the subject passes these screening procedures, then subsequent visits will involve the fat biopsies, DEXA, and other visits described below.

Fat biopsies (Visits 2, 14, 17 and 28). Regardless of the study arm assigned to all subjects will present to the CCTS fasting and a baseline fat biopsy will be performed on the thigh and lower abdomen. Abdominal and thigh subcutaneous adipose tissue will be removed by incision under local anesthesia. An ice pack will then be placed on the opposite thigh and lower abdomen for 30 min; 4 hr later, an adipose biopsy will be obtained from the iced area. The subject will then report to the CCTS daily for repeated 30 min ice pack procedures. However, at the discretion of the PI, participant may be able to perform the 30 min ice pack procedure at home. On day 7 and on day 14, subjects will report to the CCTS fasting and the above procedure will be repeated: an ice pack will be placed on the thigh and abdomen for 30 min, and fat biopsies will be taken from the iced area and from the non-iced area 4 hr later.

Propranolol Arm: Subjects who qualify for this subgroup will be given propranolol 10 mg three times per day. If they tolerate the medication well with no side effects, after 5 days, they will then increase the dose to 20 mg three times per day. If they tolerate the 20 mg dose well with no side effects, after another 5 days (day 10), they will then increase the dose to 40 mg three times per day and stay on this for the duration of the study.

Heavy Water Arm: Subjects who qualify for this subgroup will be given heavy water (at visit 2) every 3 hours for the next 12 hours while at the CCTS. They will then be sent home with doses of heavy water in sealed sterile vials, and will take one vial of heavy water twice per day for 5 weeks.

The following test and procedures will be performed on subjects:

Glucose tolerance test (Visits 1 and 15). This will be a standard oral glucose tolerance test using 75 g of glucose, with blood for glucose and insulin drawn at times 1, 30, 60, 90, and 120 min.

Resting metabolic rate. The investigator will measure resting metabolic rate (RMR). RMR is measured early in the morning, fasting, in a room on the CCTS.

DEXA. Body composition will be measured with DEXA.

12-Lead ECG: To examine heart rhythm and heart rate and any evidence of previous heart disease.

Urine Collection: Females who are capable of becoming pregnant will also be given a urine pregnancy test. If the test results show that they are pregnant they will not be able to participate in the study.

Unscheduled Visits: During the study if either the subject or the PI feel that that the subject should be seen for an additional visit due to an adverse event, the study staff will arrange for this visit. This visit should take no more than 30 minutes. During this visit the investigator will:

* Review subject's current medication use, including over the counter medications and herbals.
* Ask the subject questions about their health or any problems they may have had since their last visit.
* If necessary, take a blood sample (about 1 tablespoon) and urine sample (about 6 teaspoons) to monitor the subject's general health.
* If necessary, perform a ECG and measure blood pressure and pulse.
* If necessary, ask questions about how study drug dosing at home.

After completing the above procedure, the subject will be asked to come back for the same set of procedures the following season (i.e. winter, if original procedure was summer, or vice versa).

Therefore, if the subject completes all the procedures in both seasons, a total of 16 biopsies will be performed. Following initial studies, the investigator may refine the protocol and take fewer biopsies. For example, if early experiments determine that abdominal fat is not responsive to seasons, the investigator may discontinue this procedure. The investigator may determine that the baseline fat biopsy (prior to icing) is unnecessary.

ELIGIBILITY:
Inclusion Criteria:

* the lean subjects body mass index (BMI) < 27
* subjects with obesity/MetS (BMI 27-45 with IGT, IFG, or 3 features of MetS)
* Insulin resistance Fasting blood sugar >126, or 2 hr glu >200, but with A1C<7.5 (i.e. we will include subjects with T2DM on no meds and with good glycemic control)
* adequate platelet count (>100,000)
* hematocrit of >32
* stable weight

Exclusion Criteria:

* obese subjects (BMI > 45)
* anti-inflammatory drugs, β-blockers, any diabetes drugs or drugs known to affect adipose tissue
* an unstable medical condition
* coronary artery disease
* congestive heart failure
* heart block or a history of or any contraindication to a β-blocker.
* asthma
* previous stroke
* use of anticoagulants or aspirin
* pregnant or breastfeeding
* lifestyles involving absent or extreme temperature exposure (eg. homebound or institutionalized subjects, outdoor workers).

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-03; Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
WAT changes during repeated exposure to cold temperatures | 28 Weeks (Summer and Winter Seasons)
  Adipose biopsies will be performed
WAT changes following Propranolol dosing | 17 days in the summer season
  Subjects will be prescribed propranolol and adipose biopsies will be obtained.
In vivo measurement of adipose lipolysis and triglyceride (TG) turnover | 5 weeks per season (summer and winter)
  The heavy water will be given to and adipose biopsies will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Kern, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center Center for Clinical and Translational Science, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Finlin BS, Memetimin H, Confides AL, Kasza I, Zhu B, Vekaria HJ, Harfmann B, Jones KA, Johnson ZR, Westgate PM, Alexander CM, Sullivan PG, Dupont-Versteegden EE, Kern PA. Human adipose beiging in response to cold and mirabegron. JCI Insight. 2018 Aug 9;3(15):e121510. doi: 10.1172/jci.insight.121510. eCollection 2018 Aug 9. PMID 30089732
- [Derived] Thiagarajan D, Quadri N, Jawahar S, Zirpoli H, Del Pozo CH, Lopez-Diez R, Hasan SN, Yepuri G, Gugger PF, Finlin BS, Kern PA, Gabbay K, Schmidt AM, Ramasamy R. Aldose reductase promotes diet-induced obesity via induction of senescence in subcutaneous adipose tissue. Obesity (Silver Spring). 2022 Aug;30(8):1647-1658. doi: 10.1002/oby.23496. PMID 35894077

DOCUMENTS (1):
  • Informed Consent Form (2018-06-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT02596776/ICF_000.pdf